CLINICAL TRIAL: NCT03407703
Title: HCV Cure and Kidney Health: A Prospective, Observational Cohort Study of HCV Genotype 1 and 4 Infected Adults With and Without HIV Infection
Brief Title: Hepatitis C (HCV) Cure and Kidney Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Phyllis Tien, Professor of Medicine and Clinical Pharmacy and Staff Physician, San Francisco Veterans Affairs Medical Center
Other Study IDs: 17-22790
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C
Keywords: genotype 1; genotype 4
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma and PBMC (peripheral blood mononuclear cell)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Elbasvir / Grazoprevir Oral Tablet [Zepatier] — HCV treatment

SUMMARY:
The purpose of this study is to learn how 12 weeks of HCV treatment with elbasvir and grazoprevir (brand name Zepatier) impacts your kidney function.

DETAILED DESCRIPTION:
Prospective data collection of 25 Genotype 1 or 4 HCV-infected women from the San Francisco Women's Interagency HIV Study (WIHS) site and 25 Genotype 1 or 4 HCV-infected men from the San Francisco VA Medical Center who are initiated on Zepatier for 12 weeks (Total n=50). For women and men with HCV genotype 1a infection, only those without baseline NS5A resistance mutations will be included. Blood/urine samples will be collected before initiation of treatment, 4 weeks after treatment initiation, 12 weeks after treatment initiation (end of treatment), 24 weeks after treatment initiation to determine Sustained Virological Response (SVR), and at 48 weeks after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Active Genotype 1 or 4 HCV infection (If with Genotype 1a infection, only those without baseline NS5A resistance mutation will be included; Genotype 4 HCV infection is uncommon in both study populations). Subjects with HIV coinfection are included. We will not exclude patients who have severe Chronic Kidney Disease, are on dialysis, or have undergone kidney transplant.

Exclusion Criteria:

1. HCV genotype 2, 3, 5, or 6 infection
2. Previous virologic failure to regimens containing an NS5A inhibitor
3. Decompensated liver disease (Child-Pugh Class B or C)
4. Albumin below 3g/dL
5. Platelet count below 75,000
6. Any condition that the investigator considers a contraindication to study participation including limited life expectancy
7. Pregnant or breastfeeding woman
8. Hepatitis B virus (HBV) surface antigen positive (Note: Patients positive for the HBV core antibody will not be excluded, but will have HBV DNA levels checked and will be monitored while on Direct Acting Antivirals (DAA) therapy and medically managed as considered appropriate)
9. Documented ongoing nonadherence to prescribed medications or medical treatment, failure to complete HCV disease evaluation appointments and procedures or unable to commit to scheduled followup/monitoring for the duration of treatment
10. Poor venous access not allowing screening laboratory collection
11. Known hypersensitivity to elbasvir/grazoprevir
12. Co-administration with drugs that are 1) strong CYP3A inducers (e.g., phenytoin, carbamazepine, rifampin); 2) OATP1B1/3 inhibitors (e.g., cyclosporine, darunavir, atazanavir, tipranavir, lopinavir or saquinavir) or 3) efavirenz

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 Genotype 1 or 4 HCV-infected women from the San Francisco WIHS site and 25 Genotype 1 or 4 HCV-infected men from the San Francisco VA Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate and injury | 1 year
  measured by Cystatin C
glomerular filtration rate and injury | 1 year
  measured by Creatinine
glomerular filtration rate and injury | 1 year
  measured by albuminuria
Tubule dysfunction | 1 year
  measured by α1-microglobulin
Tubule dysfunction | 1 year
  measured by beta2-microglobulin
Tubule injury | 1 year
  measured by Interleukin-18
tubule injury | 1 year
  measured by Kidney injury molecule-1
tubule injury | 1 year
  measured by Neutrophil gelatinase-associated lipocalcin (NGAL)
tubule injury | 1 year
  measured by Clusterin
tubule injury | 1 year
  measured by Trefoil factor-3 (TFF-3)

SECONDARY OUTCOMES:
HCV clearance | 1 year
  measured by HCV viral load
liver fibrosis | 1 year
  liver stiffness measured by transient elastography

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis C Tien, MD, Principal Investigator — San Francisco VA Medical Center
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No